CLINICAL TRIAL: NCT00784420
Title: Open-Label, Randomized, 3-Way Crossover Study To Estimate The Interaction Between Multiple Dose Raltegravir And UK-453,061 In Healthy Subjects
Brief Title: Drug Interaction Study Between Raltegravir And UK-453,061
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A5271019
Record Dates: First submitted 2008-09-30; First posted 2008-11-04 (Estimated); Last update posted 2008-11-18 (Estimated); Status verified 2008-11

CONDITIONS: Healthy Volunteers
Keywords: Drug Interaction, Pharmacokinetics
MeSH Terms: interventions — UK 453,061; Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- UK-453,061 (Active Comparator)
  Interventions: Drug: UK-453,061
- Raltegravir (Active Comparator)
  Interventions: Drug: Raltegravir
- UK-453,061 plus Raltegravir (Experimental)
  Interventions: Drug: UK-453,061; Drug: Raltegravir

INTERVENTIONS:
Drug: UK-453,061 — UK-453,061 1000 mg once daily for 10 days
  Arms: UK-453,061 plus Raltegravir
Drug: UK-453,061 — UK-453,061 1000 mg once daily for 10 days
  Arms: UK-453,061
Drug: Raltegravir — Raltegravir 400 mg twice daily for 10 days
  Arms: Raltegravir
Drug: Raltegravir — Raltegravir 400 mg twice daily for 10 days
  Arms: UK-453,061 plus Raltegravir

SUMMARY:
The purpose of this study is to estimate the effect of steady state raltegravir on the steady state pharmacokinetics of UK-453,061 and steady state UK-453,061 on the steady state pharmacokinetics of raltegravir.

ELIGIBILITY:
Inclusion Criteria:

Healthy male and/or female subjects between the ages of 18 and 55 years, inclusive; Body Mass Index (BMI) of 18 to 30 kg/m2; and a total body weight >50 kg (110 lbs). A BMI lower limit of 17.5 kg/m2 may be rounded up to 18.0 kg/m2; a BMI upper limit of 30.5 kg/m2 may be rounded down to 30.0 kg/m2 and will be acceptable for inclusion.

Exclusion Criteria:

Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease; Treatment with an investigational drug within 30 days or 5 half-lives (whichever is longer) preceding the first dose of study medication; Use of tobacco- or nicotine-containing products in excess of the equivalent of 5 cigarettes per day.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2008-09; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Raltegravir plasma pharmacokinetic parameters: Cmax and AUC12 | 11 days
UK-453,061 plasma pharmacokinetic parameters: Cmax and AUC24 | 11 days

SECONDARY OUTCOMES:
Raltegravir plasma pharmacokinetic parameters: Tmax, t1/2, AUCinf, and C12h | 11 days
Safety and toleration assessed by spontaneous reporting of adverse events, vital signs, 12-lead ECG and laboratory safety assessments | 11 days
UK-453,061 plasma pharmacokinetic parameters: Tmax, t1/2, AUCinf, and C24h | 11 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5271019&StudyName=Drug%20Interaction%20Study%20Between%20Raltegravir%20And%20UK-453%2C061